CLINICAL TRIAL: NCT03358758
Title: Retrospective Morbidity and Mortality Study of Conflict-Related Injuries: Erbil, Iraq
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Maximilian Nerlander, Dr, Karolinska Institutet
Other Study IDs: 06032017
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Wounds and Injuries; War-Related Injuries; Gunshot Wound; Blast Injuries
Keywords: Trauma; War-Related Injuries; Firearm; Explosion; Bomb; Ordnance; IED; Epidemiology; Public Health
MeSH Terms: conditions — Wounds and Injuries; War-Related Injuries; Wounds, Gunshot; Blast Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective morbidity and mortality study, using routinely collected data, investigating the epidemiology of patients with conflict-related injuries presenting to a dedicated trauma hospital in Erbil, Iraq, during the campaign to liberate Mosul from ISIS.

DETAILED DESCRIPTION:
Trauma is a major cause of morbidity and mortality worldwide. An analysis of the Global Burden of Disease study indicated that in 2013, globally 973 million traumatic injuries warranted medical intervention, while 4.8 million injuries were fatal. The Small Arms Survey - Global Burden of Armed Violence report compiles worldwide conflict-related data and indicates that between 2007-2012, there were a total of 508,000 fatalities attributable to interpersonal violence worldwide, of which 70,000 were conflict-related. Since the U.S. invasion of Iraq in 2003, the country has perpetually constituted a scene of conflict. Hagopian et al reports that in the period 2003-2011, there were between 48,000 and 751,000 excess deaths attributable to the conflict.

In 2014, a new group, Islamic State of Iraq and Syria (ISIS), made significant territorial gains in several governorates in Iraq and captured key cities, including Fallujah and Mosul. ISIS is unique among terrorist groups in that it employs a combination of conventional maneuver warfare tactics with terrorist tactics such as Improvised Explosive Devices (IEDs) and Vehicle-Born Improvised Explosive Devices (VBIEDs) in order to capture and hold territory. These indiscriminate tactics lead to excessive civilian casualties.

In mid-October 2016 the offensive to liberate Mosul started. Emergency Hospital (EH) is one hospital assigned by the Kurdistan Ministry of Health to receive trauma patients from the conflict, and is located in Erbil, around 94 Km east of Mosul. EH is a dedicated trauma hospital that was set up in 1997. Since mid-October 2016 EH is exclusively providing care to injured from the armed conflict. Initially EH and WEH were the only hospitals providing surgical trauma care to patients from Mosul but since late December 2016 secondary facilities have opened closer to Mosul. The two hospitals are since then mainly referral hospitals.

Previous research on trauma from conflict zones generally focus solely on military combatants. Due to the use of ballistic protection and forward surgical teams these results may not be applicable to a civilian setting. A few organizations, such as the Médecins Sans Frontières (MSF), have reported on civilian casualties in conflict zones; however, these have been reports from single centers and articles are sometimes published several years after the trauma occurred. More timely information is needed on the type and pattern of injury for both combatants and civilians. ISIS tactics are likely to have a significant impact on the type of injuries seen at EH. An increased understanding of this impact is essential for addressing emerging resource requirements. The investigators anticipate a high incidence of blast- and firearm-related injuries in both civilians and combatants. This study utilizes existing data from the hospital to gain knowledge of the characteristics of conflict-related injuries, as well as the demographic profile of the patients. Furthermore, the data will be used to investigate how morbidity and mortality varies depending on injury type.

Specific aims:

1. Describe the demographics of patients with conflict-related injuries presenting to the EMC during the Mosul campaign.
2. Describe the morbidity profile of the study population, specifically:

   1. Determine how markers for injury severity vary with injury mechanism and patient status as combatant or non-combatant.
   2. Compare how injury mechanism varies with patient identity as non-combatant, ISF or Peshmerga.
3. Determine the in-hospital mortality rate.

This is essential both for generating actionable results necessary to direct operational priorities, and gaining an understanding of the wider public health impact of the ongoing conflict. The evidence generated by this study will facilitate effective programmatic monitoring and help optimize resource allocation to meet the rapidly changing health needs in the area.

ELIGIBILITY:
Inclusion criteria: All patients from Mosul presenting with conflict-related injuries to Emergency Hospital between October 16, 2016 to July 10, 2017.

-

Exclusion Criteria:

* Non-conflict related injures, Patients not categorised as either civilian or combatant

Max Age: 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Civilians and combatants injured in Mosul
Sampling Method: Non-Probability Sample
Enrollment: 1832 (Actual)
Dates: Start 2016-10-16 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Morbidity | October 16, 2016 to July 10, 2017
  Site of injury, mechanism of injury, patient status as combatant or non-combatant
Mortality | October 16, 2016 to July 10, 2017
  In-hospital mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institute, Stockholm, Sweden

REFERENCES:
- [Derived] Nerlander MP, Haweizy RM, Wahab MA, Alga A, von Schreeb J. Epidemiology of Trauma Patients from the Mosul Offensive, 2016-2017: Results from a Dedicated Trauma Center in Erbil, Iraqi Kurdistan. World J Surg. 2019 Feb;43(2):368-373. doi: 10.1007/s00268-018-4817-1. PMID 30357467